CLINICAL TRIAL: NCT03762135
Title: Location Initiated Individualized Texts for Adolescent Health (LIITAH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Susan J Woolford, MD, MPH, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM0000143430; 2R42MD008840-02 (NIH)
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Overweight; Obese; Healthy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full version of the LIITah App. (Experimental): Participants will be given the LIITAH app. which consists of 1) enhanced location identification (ELI), 2) self reported nutrients by annotated photos (SNAP), 3) delivery of individually and culturally tailored point of purchase (POP) prompts along with tailored messages sent at other times of the day, 4) use of app. in connection with parents, 5) goal setting, 6) a point system
  Interventions: Other: Full version of the LIITah App.
- Partial App. (ELI and SNAP only) (Active Comparator): Participants will be given only the ELI and SNAP components. It will detect their presence in a restaurant and allow users to document their purchases by submitting annotated photos, but it will not deliver any POP prompts encouraging them to make healthy choices, or messages at other times of the day.
  Interventions: Other: Partial App. (ELI and SNAP only)

INTERVENTIONS:
Other: Full version of the LIITah App. — Participants will download the LIITAH app. For the first 2 weeks the app. will only record presence in a restaurant and ask users to submit photos of their food. in week 3 all of the program features will be activated.
  Arms: Full version of the LIITah App.
Other: Partial App. (ELI and SNAP only) — Participants will download the LIITAH app. It will detect their presence in a restaurant and users will submit annotated photos of their purchases
  Arms: Partial App. (ELI and SNAP only)

SUMMARY:
The goal of this study is to test whether the mobile application (app.) helps adolescents make healthy food choices, decreasing calories purchased from restaurants, fewer number of visits to restaurants, and if it has an impact on their body mass index (BMI). Eligible adolescents will be enrolled in the study along with a parent for approximately 6 weeks.

DETAILED DESCRIPTION:
Excess weight puts millions of adolescents in the US at risk for weight-related illnesses and premature death and disproportionately impacts Black and Hispanic populations. Black and Hispanic youth are more likely to be exposed to communities with high densities of fast-food restaurants. This project sought to help adolescents make healthy choices in obesogenic settings that are relevant to and have been tested in populations who are at the highest risk for obesity and its associated costs.

Previous research revealed that adolescents welcomed health-related text messages (based on Self Determination Theory and Motivational Interviewing) if they viewed them as personally relevant and if they were received at times when they faced dietary choices. Based on these findings, the following is hypothesized: delivering messages (tailored to users' preferences and values) at a time and place when they are making a dietary choice (e.g., in a restaurant) will positively influence their choices.

Thus, the Health Kick+ App was developed, and it aimed to deliver tailored messages at the point of purchase. This app identifies when users are in a restaurant, automatically sends culturally relevant messages tailored to user preferences and the menu options at their location with the aim of prompting users to make a healthy choice, and allows users to submit an annotated photo response about their food choice. Participants were recruited as parent/guardian and teen dyads. Teen participants also were allowed to set goals, see progress reports, and receive daily health tips. Parent/guardian participants could communicate with the teen via the app and monitor progress.

This project worked towards enhancing the earlier version of the app developed in the LIITA3H study. The LIITAH study worked towards developing 1) deeper individual tailoring, making the content even more relevant to users from different races/ethnicities; 2) a dyad capability for parents to use the app coordinated with their adolescent; and 3) additional engagement features to remind participants to use the app frequently.

As of 2020, due to the influence of the public health emergency, lockdowns prevented any participants from engaging in going to restaurants as they previously would have. Due to the trial beginning in 2021, no six-month app-based data was acquired before the lockdown, and research limitations were imposed. When behavioral research of this type was allowed to resume, limited time remained before the funded study would have to end. Thus, certain aspects of the protocol and intervention were modified. To be pragmatic under these constrained circumstances, the intervention was shortened from 6 months to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* eat restaurant food at least 3 times a week and have a parent who agrees to participate.

Exclusion Criteria:

-

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Woolford, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 78 parents were also consented on behalf of their children and were interviewed after data was collected for their child for qualitative, non-health-outcome related measures. Therefore, they are not included as an arm as no intervention was received.
Period: Overall Study
Arm/Group | Full Version of the LIITah App. | Partial App. (ELI and SNAP Only)
Started (Started represents 78 dyads (78 parents of 78 adolescents) who consented, downloaded the apps, and began participation.) | 52 (Participant flow is based on dyads of 1 parent and 1 adolescent.) | 26 (Participant flow is based on dyads of 1 parent and 1 adolescent.)
Completed | 52 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: With the exception of region of enrollment, baseline data shown are for the adolescent participants only because no age, BMI, or other baseline data shown in baseline characteristics were collected from parents. Region of enrollment data was available for parents because all parents in dyads were co-located with their children who were the object of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Version of the LIITah App. | Partial App. (ELI and SNAP Only) | Total
Number analyzed (Participants) | 52 | 26 | 78
Age, Continuous [Mean (Full Range); unit: years] | 15 [13 to 17] | 15 [13 to 17] | 15 [13 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 15 | 53
  Male | 14 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 33 | 17 | 50
  More than one race | 7 | 3 | 10
  Unknown or Not Reported | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Middle Eastern | 1 | 0 | 1
  Not Hispanic, Latino, or Middle Eastern | 45 | 24 | 69
Region of Enrollment [Count of Participants; unit: Participants] — Adolescent participant data only
  Participants
    United States | 52 | 26 | 78
Region of Enrollment [Number; unit: parents of participants] — Parents
  parents of participants
    United States | 52 | 26 | 78
Estimated number of fast food restaurant visits per week prior to study [Mean (Full Range); unit: FFR Visits] | 5 [3 to 10] | 5 [3 to 12] | 5 [3 to 12]
BMI Percentile [Mean (Full Range); unit: BMI (kg/m^2) Percentile] | 87.2 [52.9 to 99.9] | 87.4 [65.7 to 99.7] | 87.3 [52.9 to 99.9]
Ethnic Identity Score [Mean (Full Range); unit: units on a scale] — The Ethnic Identity Score (Multigroup Ethnic Identity Measure) is an instrument assessing affiliation and identification with one's ethnic group. Scores range from 1 (least identified) to 4 (most identified). Only participants who identified as African American, Hispanic, or multiple races including African American were administered this survey. Population: Only participants who identified as African American, Hispanic, or multiple races including African American were administered this survey.
  units on a scale
    number analyzed (Participants) | 21 | 8 | 29
    (all) | 3.2 [2.3 to 3.8] | 3.0 [2.2 to 3.6] | 3.2 [2.2 to 3.8]

OUTCOME MEASURES:

1. Primary Outcome: Visits to Restaurants
Description: Number of visits will be obtained from the app. This outcome measure is based exclusively on adolescent data.
Time Frame: over 6 weeks
Measure: Mean (Standard Deviation); unit: Number of FFR Visits
Arm/Group | Full Version of the LIITah App. | Partial App. (ELI and SNAP Only)
Number analyzed (Participants) | 52 | 26
Number of FFR Visits
  Week 1 | 3.1 (3) | 2.6 (2)
  Week 2 | 2.9 (2.6) | 2.6 (2.1)
  Week 3 | 2.5 (2.3) | 2.1 (1.5)
  Week 4 | 1.9 (2.1) | 2.1 (1.3)
  Week 5 | 2 (2.1) | 1.7 (1.7)
  Week 6 | 1.6 (1.7) | 1.6 (1)

2. Primary Outcome: Calories Purchased From Restaurants
Description: Number of calories purchased by the adolescent and for the adolescent were assessed using annotated photos, and nutritional data from the restaurant menus.
  This analysis used population averaged generalized estimating equation regressions (GEE) to compare trajectories of calories purchased between groups. The GEE approach allowed for the correlation in repeated observations collected from participants over time. This outcome measure is based exclusively on adolescent data.
Time Frame: over 6 weeks
Measure: Mean (95% Confidence Interval); unit: Calories
Arm/Group | Full Version of the LIITah App. | Partial App. (ELI and SNAP Only)
Number analyzed (Participants) | 52 | 26
Calories
  Week 1 | 2432 [1927 to 2936] | 2035 [1570 to 2500]
  Week 2 | 2162 [1740 to 2583] | 1982 [1611 to 2352]
  Week 3 | 1892 [1531 to 2252] | 1929 [1584 to 2274]
  Week 4 | 1622 [1288 to 1955] | 1876 [1475 to 2277]
  Week 5 | 1352 [1002 to 1701] | 1823 [1310 to 2335]
  Week 6 | 1082 [679 to 1484] | 1769 [1117 to 2422]
Statistical Analysis 1: Comparison: Full Version of the LIITah App. vs Partial App. (ELI and SNAP Only); Test type: Superiority; p = 0.044, GEE Linear Regression — This relates to the entirety of the 6-week period; Generalized Estimation Equation Linear Regression

3. Secondary Outcome: Body Mass Index (BMI) Percentile
Description: Height and weight will be obtained. This outcome measure is based exclusively on adolescent data.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: BMI (kg/m2) percentile
Arm/Group | Full Version of the LIITah App. | Partial App. (ELI and SNAP Only)
Number analyzed (Participants) | 52 | 26
BMI (kg/m2) percentile | 85.4 [48.7 to 99.9] | 88.1 [47.4 to 99.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from each adolescent's initial enrollment to their last interview; the interval between these events for each participant was typically 6 weeks.
Description: Parents did not receive the intervention. No adverse event data was collected from parents.
Groups:
- Full Version of the LIITah App. (Adolescents): Participants will be given the LIITAH app. which consists of 1) enhanced location identification (ELI), 2) self reported nutrients by annotated photos (SNAP), 3) delivery of individually and culturally tailored point of purchase (POP) prompts along with tailored messages sent at other times of the day, 4) use of app. in connection with parents, 5) goal setting, 6) a point system
  Full version of the LIITah App.: Participants will download the LIITAH app. For the first 2 weeks the app. will only record presence in a restaurant and ask users to submit photos of their food. in week 3 all of the program features will be activated.
- Full Version of the LIITah App.(Parents): Parents of adolescents who received the LIITAH app.
- Partial App. (ELI and SNAP Only) (Adolescents): Participants will be given only the ELI and SNAP components. It will detect their presence in a restaurant and allow users to document their purchases by submitting annotated photos, but it will not deliver any POP prompts encouraging them to make healthy choices, or messages at other times of the day.
  Partial App. (ELI and SNAP only): Participants will download the LIITAH app. It will detect their presence in a restaurant and users will submit annotated photos of their purchases
- Partial App. (ELI and SNAP Only) - Parents: Parents of adolescents who received the ELI and SNAP components.
Arm/Group | Full Version of the LIITah App. (Adolescents) | Full Version of the LIITah App.(Parents) | Partial App. (ELI and SNAP Only) (Adolescents) | Partial App. (ELI and SNAP Only) - Parents
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/26 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/26 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT03762135/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT03762135/ICF_000.pdf